CLINICAL TRIAL: NCT06952894
Title: Feasibility and Efficacy of Surgical Navigation 'RUS Lung' in Patients Undergoing Minimally Invasive Thoracic Surgery (MITS) Segmentectomy for Lung Cancer: a Multicenter Prospective Observational Study With a Propensity-score Matching Analysis
Brief Title: Feasibility of RUS Lung in MITS
Acronym: HTL-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hutom Corp (Industry)
Collaborators: Severance Hospital (Other); Ajou University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTL-001
Record Dates: First submitted 2025-04-09; First posted 2025-05-01 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: lung cancer; 3D model; 3 dimensional; segmentectomy; robot-assisted thoracoscopic surgery; video-assisted thoracoscopic surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RUS Group (Experimental): Patients undergo video-assisted or robot-assisted thoracoscopic surgery using RUS Lung software.
  Interventions: Device: RUS Lung

INTERVENTIONS:
Device: RUS Lung — The RUS Lung is an endoscopic imaging treatment planning software program. It creates a patient-specific simulation of the thoracic surgical environments, allowing for the visualization of tumor, bronchovascular structures and thoracic organs during the surgical planning process and the operation. RUS Lung utilizes preoperative CT images of the patients to segment tumor, organs, blood vessels, and bronchus and reconstructs them into a 3D model. Although there is no direct intervention on the patient, the surgeon uses RUS Lung as a surgical navigation tool to simulate the surgery before performing the actual procedure.

SUMMARY:
This sponsor-initiated prospective observational study aims to demonstrate the feasibility and efficacy of RUS Lung Surgical Navigation System in patients undergoing minimally invasive thoracic surgery(MITS). The trial will enroll 36 patients who undergo video-assisted or robot-assisted thoracoscopic surgery using RUS Lung. The study will be conducted across two medical centers."

* Investigational Medical Device: RUS Lung (Endoscopic Imaging Treatment Planning Software)
* Clinical Trial duration: 12 months from IRB approval
* Target number of subjects: Total of 36 participants

DETAILED DESCRIPTION:
Patients will be enrolled after being selected based on the inclusion and exclusion criteria and after obtaining informed consent. Video-assisted or robot-assisted thoracic surgery (VATS/RATS) will be performed using RUS Lung.Parameters-associated with operation or clinical outcomes will be evaluated during hospitalization period or through outpatient follow-ups for up to 2 weeks after discharge. The operative outcomes including operative time, estimated blood loss, complication rates, and hospital length were compared with the historical control underwent VATS and RATS without using RUS Lung.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed with lung caner (tumor size≤3cm)
* Individuals aged 19 or older
* Individuals who who are able to undergo CT imaging according to the established protocol
* Individuals who have voluntarily given written consent to participate in this clinical trial

Exclusion Criteria:

* Vulnerable subjects
* Individuals who who are not able to undergo CT imaging according to the established protocol
* Individuals who are expected to have severe adhesions
* Individuals who are unable to follow the study procedures and are deemed inappropriate for participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
The concordance rate of tumor location across CT, RUS Lung, and surgery | The operative day (operative day ± 5 days)
  Overall feasibility of the RUS Lung system will be evaluated by 3 factors as below.
  1. CT turn-around time: the duration between uploading of preoperative CT and downloading the 3D model file
  2. The stability of the RUS Lung system
  3. The concordance rate of tumor location across CT, RUS Lung, and surgery

SECONDARY OUTCOMES:
The degree of consistency between surgical planning using the RUS lung system and actual surgical findings. | From enrollment to the end of treatment at 2 weeks
  1. The consistency of surgical planning (using CT and RUS, respectively) and operative findings
  2. Surgical outcomes (operative time, estimated blood loss, hospital length, and complication rates)
  3. User convenience

CONTACTS AND LOCATIONS:
Overall Officials: Chang Young Lee, M.D.,Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided